CLINICAL TRIAL: NCT04254835
Title: Assessment of Inhibition of Biofilm Formation and Plaque Bacterial Count of Fluoride Varnish Containing Chlorhexidine and Cetylpyridinium Chloride Versus Conventional Fluoride Varnish Among High Caries Risk Patients: Randomized Clinical Trial
Brief Title: Assessment of Inhibition of Biofilm Formation and Plaque Bacterial Count of Fluoride Varnish Containing Chlorhexidine and Cetylpyridinium Chloride Versus Conventional Fluoride Varnish
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Hesham Mohamed, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 221091
Record Dates: First submitted 2019-07-15; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: High Caries Risk Patients
MeSH Terms: interventions — Fluor Protector

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): Varnish containing Fluoride, Chlorhexidine and Cetylpyridinium Chloride (Cervitec F, Ivoclar Vivadent - Schaan Liechtenstein) will applied to this group once at the beginning of the study.Plaque and bacterial count will be evaluated at intervals 2 weeks,4 weeks,12 weeks, and 24 weeks.
  Interventions: Drug: Cervitec F, Ivoclar Vivadent - Schaan Liechtenstein
- control group (Active Comparator): Varnish containing Fluoride (Fluor Protector, Ivoclar Vivadent - Schaan Liechtenstein). will applied to this group once at the beginning of the study.
  Plaque and bacterial count will be evaluated at intervals 2 weeks,4 weeks,12 weeks, and 24 weeks.
  Interventions: Drug: Fluor Protector, Ivoclar Vivadent - Schaan Liechtenstein

INTERVENTIONS:
Drug: Cervitec F, Ivoclar Vivadent - Schaan Liechtenstein — Fluoride varnish containing Chlorhexidine and Cetylpyridinium Chloride
  Arms: intervention group
Drug: Fluor Protector, Ivoclar Vivadent - Schaan Liechtenstein — Conventional Fluoride varnish
  Arms: control group

SUMMARY:
Two different Fluoride varnish systems(Fluoride varnish containing Chlorhexidine and Cetylpyridinium Chloride (CPC) and conventional fluoride) will be applied to high caries risk patients to assess their clinical effects on plaque accumulation and plaque bacterial count .

DETAILED DESCRIPTION:
Preoperative steps:

* The diagnostic chart will be filled including all data about the patient's medical history, dental history, plaque assessment and plaque bacterial count.
* Scaling and polishing will be carried out for subjects.

clinical steps:

* Control Group: Conventional Fluoride varnish (Fluor Protector, Ivoclar Vivadent - Schaan Liechtenstein) will be applied on dry teeth in a thin layer, allowed to dry for 1 minute, and participants will be instructed to avoid rinsing after application, only spitting. Eating, drinking and brushing should be avoided for 1 hour after varnish application.
* Intervention Group: Varnish containing Fluoride, Chlorhexidine and Cetylpyridinium Chloride (Cervitec F, Ivoclar Vivadent - Schaan Liechtenstein) will be applied on dry teeth in a thin layer, allowed to dry for 1 minute, and participants will be instructed to avoid rinsing after application, only spitting. Eating, drinking and brushing should be avoided for 1 hour after varnish application.

Each participant will be assessed for plaque retention using plaque index and Standardized photography and image analysis to disclosed dental plaque, and plaque bacterial count using culture media sensitive for mutans streptococci (MS) in the following intervals:

* Enrolment Baseline assessment
* First visit (2nd week)
* Second visit (4th week)
* Third visit (12th week)
* Fourth visit (24th week)

ELIGIBILITY:
Inclusion Criteria:

Patients with good general state of health.

* No signs of periodontitis.
* Patients had a recorded high bacterial count after caries risk assessment.
* No antibiotic treatment within 1 month prior to the start of the trial.
* No current medication with anti-inflammatory drugs.
* No use of antiseptic mouth rinses.
* Non-smokers.

Exclusion Criteria:

* Patients with disabilities, systemic disease or severe medical conditions.

  * Patients with severe or active periodontal disease.
  * Antibiotic treatment within 1 month prior to the start of the trial.
  * Current medication with anti-inflammatory drugs.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Plaque Retention | Patient will be evaluated at 2nd week of the study in the morning before teeth brushing.
  Checked using a disclosing agent by Silness and Löe Dental Plaque index
Plaque Retention | Patient will be evaluated at 4th week of the study in the morning before teeth brushing.
  Checked using a disclosing agent by Silness and Löe Dental Plaque index
Plaque Retention | Patient will be evaluated at 12th week of the study in the morning before teeth brushing.
  Checked using a disclosing agent by Silness and Löe Dental Plaque index
Plaque Retention | Patient will be evaluated at 24th week of the study in the morning before teeth brushing.
  Checked using a disclosing agent by Silness and Löe Dental Plaque index

OTHER OUTCOMES:
Plaque bacterial count | Patient will be evaluated at 2nd, 4th, 12th and 24th week of the study in the morning before teeth brushing.
  Culture media for mutans streptococci (MS) is used to measure (MS) count in collected plaque samples

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry Cairo Universty, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No